CLINICAL TRIAL: NCT01249846
Title: The Efficacy and Safety of 2.5 mg Chlorhexidine Gluconate Chip (PerioChip®) in Frequent Treatment Versus Routine Treatment in Therapy of Adult Chronic Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Dr. Avi Avramoff, V.P R&D, Dexcel Pharma Technologies Ltd.
Purpose: Treatment
Other Study IDs: CLI/015P
Record Dates: First submitted 2010-11-28; First posted 2010-11-30 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Generalized Adult Periodontitis
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Each one of the two selected periodontal pockets (target pockets) will be randomized to the Frequent PerioChip® treatment or to the Routine PerioChip®.
  Interventions: Drug: PerioChip ®
- Arm 2 (Placebo Comparator): Each one of the two selected target pockets will be randomized to the Frequent PerioChip® treatment or to the Frequent Placebo Chip treatment.
  Interventions: Drug: PerioChip ®

INTERVENTIONS:
Drug: PerioChip ®

SUMMARY:
The purpose of this study is to assess the efficacy and the safety of Chlorhexidine Gluconate Chip (PerioChip®) in frequent treatment versus routine treatment in therapy of adult chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form.
2. Good general health.
3. Male or female patients aged >21 years old.
4. Availability for the 25 week duration of the study.
5. Chronic periodontal disease on natural teeth
6. Females of childbearing potential must be non-pregnant and non-lactating at entry and agree to use an adequate method of birth control during the study.

Exclusion Criteria:

1. Oral health or factor that may influence the outcome of the study.
2. History of allergy to Chlorhexidine .
3. Patient uses Chlorhexidine oral rinses/mouthwashes on a regular basis.
4. Patients treated with medications that may influence the outcome of the study.
5. Presence of any of the following conditions: Type 1 diabetes, un-controlled type II diabetes, major recurrent aphtae stomatitis, abscesses and related oral pathologies.
6. The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
7. Patient participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, School of Graduate Dentistry, Rambam Health Care Center, Haifa, Israel